CLINICAL TRIAL: NCT02850575
Title: Etude Prospective, Multicentrique, Non contrôlée, Non randomisée, Ouverte Pour l'évaluation de la Fixation Osseuse d'Une Cupule hémisphérique, le Mpact® Double Mobilité
Brief Title: Bone Fixation of Mpact Double Mobility Cup
Status: Active, not recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.017.01
Record Dates: First submitted 2016-07-22; First posted 2016-08-01 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Total Hip Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Mpact Double Mobility cup

SUMMARY:
This study aims to evaluate long term fixation of the Mpact Double Mobility cup trough IMAGIKA technology.

ELIGIBILITY:
Inclusion Criteria:

* primary hip replacement
* patients 18 to 80 years old
* patients who accept the follow-up schedule

Exclusion Criteria:

* femoral neck fracture
* patients requiring grafts
* progressive local or systemic infections
* patients presenting muscular deficiency, neuromuscular disease or vascular insufficiency of the involved limb
* patients suffering from diseases that can compromize the recovery to independent mobility
* patients with BMI > 40
* patients with cognitive diseases that can compromize their participation in the study
* patients living in geographical area not allowing the clinical follow-up to be performed
* patients participating in other biomedical research
* patients <18 years old
* patients > 80 years old
* pregnant or breast feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible for a total hip replacement at the investigational sites will be invited in the study
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-01; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
implant fixation trough IMAGIKA | 10 years
  implant fixation trough IMAGIKA

SECONDARY OUTCOMES:
Harris Hip Score | preop, 3 months, 1, 2, 5, 10 years
  Harris Hip Score
complications | intraop, immediate postop, 3 months, 1, 2, 5, 10 years
  complications
penetration of femoral head in the polyethylene insert trough IMAGIKA | 3 months, 5 and 10 years
  penetration of femoral head in the polyethylene insert trough IMAGIKA
implant stability trough standard x-ray | 3 months, 1, 2, 5, 10 years
  implant stability trough standard x-ray
implant survival trough Kaplan-Meier curve | 3 months, 1, 2, 5, 10 years
  implant survival trough Kaplan-Meier curve
implant fixation trough IMAGIKA | 3 months and 5 years
  implant fixation trough IMAGIKA

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Générale, Annecy, France
  - Orthéo - Espace Fauriel, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No